CLINICAL TRIAL: NCT06361628
Title: Implementation and Evaluation of Tailored Interventions to Increase MMR and/or HPV Vaccine Uptake in Underserved Communities in Greece, The Netherlands, Poland and Slovakia
Brief Title: Implementation and Evaluation of Tailored Interventions to Increase MMR and/or HPV Vaccine
Acronym: RIVER-EU
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Collaborators: Prolepsis Institute for Preventive, Environmental and Occupational Medicine (Other); University in Zielona Góra (Other); Pavol Jozef Safarik University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: RIVER-EU WP4
Record Dates: First submitted 2024-03-20; First posted 2024-04-12 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Vaccination; Health Systems; Knowledge, Attitudes, Practice
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Educational sessions delivered by health promotors in Greece (Experimental): In this approach, medical professionals and health promoters-trusted members of the community-will educate refugee and migrant parents. The focus is on enhancing awareness of HPV/MMR and fostering a greater willingness to vaccinate their children/adolescents. Multicultural schools and migrant associations are the locations where the educational sessions will be provided.
  Interventions: Behavioral: multicomponent intervention on vaccination awareness
- Educational sessions delivered by health promotors and healthcare professionals in the Netherlands (Experimental): Trusted community health members will be trained and will act as health promotors in the intervention. Together with health care professionals they will offer educational sessions on HPV vaccination at locations close to where people live (in the neighborhoods) and locations communities are familiar with, such as community centers, schools, health centers, religious places or offices of foundations/non-governmental organizations. Together with local stakeholders it will be verified that locations are also acceptable for the target communities. A navigation component is also included and participants will be contacted 1 week and 3 months after the educational sessions and reminded to get vaccinated and will be asked if they still have questions or need help to find their way to get vaccinated.
  Interventions: Behavioral: multicomponent intervention on vaccination awareness
- Educational sessions delivered by health promotors in Poland (Experimental): This intervention is based on the principle of face-to-face and online health education, where Ukrainian parents are educated by general practitioners to raise HPV/MMR awareness and increase willingness to child/adolescent vaccination.
  Interventions: Behavioral: multicomponent intervention on vaccination awareness
- Educational sessions delivered by health promotors in Slovakia (Experimental): Roma health mediators will be trained on HPV vaccination and thereafter will offer educational sessions to the underserved communities. Educational sessions take place at either municipalities, schools, community centers, local health care providers and public health authorities.
  Interventions: Behavioral: multicomponent intervention on vaccination awareness

INTERVENTIONS:
Behavioral: multicomponent intervention on vaccination awareness — Educational sessions to create awareness on HPV and MMR (were addressed) vaccination that is culturally sensitive health information and provided in an easily understandable manner by trained health promoters (and healthcare professionals) to underserved communities. Support for navigation and access to vaccines.

SUMMARY:
The goal of the study is to monitor and evaluate the implementation of interventions that aim to increase HPV & MMR vaccines among underserved communities across four European countries: Greece, Netherlands, Poland, and Slovakia. The interventions will target identified health systems barriers in an earlier phase of the project. The interventions that will be implemented employ trusted community members as health promotors whom will provide educational sessions on HPV and MMR vaccination to the target groups. In addition, the cost-effectiveness of vaccine uptake strategies for the target groups is being evaluated.

The main research question is: to what extent is the multicomponent tailored intervention effective to increase MMR/HPV intention and vaccine uptake in the target population in Greece, Netherlands, Poland and Slovakia?

DETAILED DESCRIPTION:
The general objective of the study is to improve access to vaccination by addressing relevant system level barriers to increase HPV and MMR (where applicable) vaccine intention and uptake among the target groups. The investigators expect that the intervention will address health system barriers to improve increase in access to information on vaccination and vaccination services.

A prospective multicomponent intervention study will be performed between 1st of April 2024 and 31st of July 2025 that will be evaluated using a pre and post design as well as a participatory approach during the implementation. As part of the multicomponent intervention a preparatory phase is taken place before this period of time. The multicomponent intervention consists of training of health promotors and healthcare professionals, and of educational sessions to community members and navigation. The educational sessions will be offered at suitable and accessible locations for the target population.

The five communities targeted in are the following:

1. The migrant community in Greece (HPV and MMR)
2. Turkish and Moroccan women in the Netherlands (HPV)
3. The Ukrainian community in Poland (HPV and MMR)
4. The Roma community in Slovakia (HPV)

ELIGIBILITY:
Inclusion Criteria:

* parents of children eligible for MMR and/or HPV vaccination according to country guidelines on those specific vaccines

Exclusion Criteria:

* respondents not willing or able to fill out questionnaires

Ages: 12 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Intention to vaccinate MMR and/or HPV by questionnaire | Pre and immediately following the intervention and 6 month post intervention
  Intention for vaccination against MMR and/or HPV among the underserved communities

SECONDARY OUTCOMES:
Uptake of MMR and/or HPV vaccinations by questionnaire | Pre and 6 month post intervention evaluation is necessary
  MMR and/or HPV vaccination uptake among the underserved communities
Knowledge concerning MMR and/or HPV vaccinations in the target group using a questionnaire | Pre and immediately following the intervention and 6 month post intervention evaluation
  Knowledge concerning MMR and/or HPV vaccinations among the target group
Communication skills of health care professionals using a questionnaire | Pre intervention and directly post intervention
  Communication skills of healthcare professionals to deliver appropriate information
Satisfaction of the stakeholders as measured by a questionnaire | Directly post intervention
  Satisfaction of stakeholders (health promotors and health professionals) with the implementation process and the intervention itself

OTHER OUTCOMES:
Improved access to vaccinations by addressing identified health system barriers - number of barriers addressed | Through study completion, an average of 1 year
  Addressed health system barriers to improve access to MMR and/or HPV vaccinations among the underserved communities

CONTACTS AND LOCATIONS:
Overall Officials: Nikole Papaevgeniou, PhD, Principal Investigator — Prolepsis Institute for Preventive, Environmental and Occupational Medicine; Daniela Fiľakovská, PhD, Principal Investigator — UPJS; Maria Ganczak, MD PhD, Principal Investigator — University Zielona Gora; Michael Edelstein, MD PhD, Principal Investigator — Bar Ilan University; Cornelis Boersma, PhD, Principal Investigator — University Medical Center Groningen
Locations (4):
- Prolepsis, Athens, Athene, Greece
- University Medical Center Groningen, Groningen, Netherlands
- University of Zielona Gora, Zielona Góra, Lubusz Voivodeship, Poland
- PJ Šafárik University, Košice, Košice Region, Slovakia

IPD SHARING:
Plan to Share IPD: Yes
Sharing according to the European Union open research guidelines.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: After study completion
Access Criteria: As per open research protocol - on request to principal investigator University Medical Center Groningen
URL: https://river-eu.org/